CLINICAL TRIAL: NCT04845243
Title: Compared Effectiveness of a Short Computer-based Emotion Recognition Training in Conduct Disorder and Autistic Spectrum Disorder Patients
Brief Title: Effectiveness of a Short Computer-based Emotion Recognition Training in Different Patient Groups
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Christina Stadler (Network)
Responsible Party: Sponsor-Investigator, Prof. Christina Stadler, Head Psychologist, Clinical Professor, Clinic for Children and Adolescents, University Psychiatric Clinics Basel
Organization: University Psychiatric Clinics Basel (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EmoRecTraining_EVA
Record Dates: First submitted 2021-04-08; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Autism Spectrum Disorder; Conduct Disorder
Keywords: Autism Spectrum Disorder; Emotion recognition training
MeSH Terms: conditions — Autism Spectrum Disorder; Conduct Disorder

STUDY DESIGN:
Intervention Model Description: Participants will receive six sessions (duration approx. 1h/session) of the software-based training program "Emotionen Verstehen und Ausdrücken" (EVA; Moebert & Lucke, 2019). Sessions will be administered 2-3 times/week depending on the participants' time availability. In order to objectively identify the potential benefit of the training for each participant, they will perform two separate tasks before and after the emotion recognition training, the Geneva Emotion Recognition test (GERT; Schlegel, Grandjean,& Scherer, 2014) and a social decision-making task. A comparison of their performance pre- and post-training is taken as an indicator of improvement in emotion recognition skills.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotion recognition training (Other): All participants have to complete the online emotion recognition training E.V.A. as well as the pre- and post training tasks: GERT and social decision making task.
  Interventions: Behavioral: Emotionen Verstehen und Ausdrücken (E.V.A.)

INTERVENTIONS:
Behavioral: Emotionen Verstehen und Ausdrücken (E.V.A.) — The online training is focused on the strengthening of socioemotional competences and consists of different training tasks (up to 3 million) presented to the participant as mini games. These training tasks are specifically designed according to empirical findings to match the socio-emotional recognition needs of people with ASD. During these games, an adapted Elo-Algorithm allows to automatically evaluate the participants' performance and adapts the difficulty levels throughout the users' progress in the training.

SUMMARY:
Emotion recognition and regulation are necessary skills for social interaction. Disrupted development of these processes severely interferes with socio-emotional development. These difficulties are commonly reported in patients with Autistic Spectrum Disorder (ASD) or Conduct Disorder (CD), with the subsequent social/interpersonal difficulties. The available evidence suggest that impaired emotion regulation processes might underlie the aggressive behaviours frequently observed in both disorders. However, no study has yet investigated the presence of disorder-specific characteristics on emotion processing between these two disorders. Different impaired emotion recognition difficulties may underlie the reported emotion dysregulation. A practical implication of this is that given that both disorders have shown difficulties during emotion recognition processes, a short, computer-based intervention to improve emotion recognition might benefit both cases, even though their aetiologies might differ.

DETAILED DESCRIPTION:
For ASD patients, studies training facial emotion recognition have focused on increasing the active attention to the eye region, re-directing attention to facial features to facilitate facial emotion recognition. Evidence shows positive results using computer-based emotion recognition training programs with young children and adolescents with ASD. It has also been recently suggested that emotion recognition training may be a suitable intervention for patients with CD. This would be supported by some preliminary evidence in patients with severe behavioural problems, young offenders and patients with CD + CU Traits. The overall goal of this project is to investigate the compared impact of an emotion recognition training in patients with ASD or CD. This goal can be subdivided into three separate subgoals: a) identify whether the training program is effective; b) identify whether the training program has differentiated or comparable effects between both patients groups and c) investigate individual characteristics that may help identify those individuals who would benefit most from the intervention. This information is crucial to inform the design of more efficient treatments to differentially address the specific deficits associated to the disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: ASD or CD
* German speaking
* IQ > 70
* Age: 10-18

Exclusion Criteria:

* Comorbid Anxiety or Depressive disorder diagnosis
* IQ < 70
* Insufficient German language skills
* Severe developmental disorders

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in performance accuracy in Geneva Emotion Recognition Test (GERT) | Change in performance before and after the emotion recognition training, after 1 month (pre/post measure)
  Percentage of accuracy to stimuli showing facial emotions
Change in performance response times in Geneva Emotion Recognition Test (GERT) | Change in performance before and after the emotion recognition training, after 1 month (pre/post measure)
  Response times to stimuli showing facial emotions
Change in performance reaction times in Social decision-making task | Change in Performance before and after the emotion recognition training, after 1 month (pre/post measure)
  Reaction times for each of the facial emotions shown
Change in choices in Social decision-making task | Change in choices before and after the emotion recognition training, after 1 month (pre/post measure)
  The proportion of choices that maximise their self-gain for each of the facial emotions shown

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed SP, Bittencourt-Hewitt A, Sebastian CL. Neurocognitive bases of emotion regulation development in adolescence. Dev Cogn Neurosci. 2015 Oct;15:11-25. doi: 10.1016/j.dcn.2015.07.006. Epub 2015 Jul 29. PMID 26340451
- [Background] Blakemore SJ. The social brain in adolescence. Nat Rev Neurosci. 2008 Apr;9(4):267-77. doi: 10.1038/nrn2353. PMID 18354399
- [Background] Somerville LH, Casey BJ. Developmental neurobiology of cognitive control and motivational systems. Curr Opin Neurobiol. 2010 Apr;20(2):236-41. doi: 10.1016/j.conb.2010.01.006. Epub 2010 Feb 16. PMID 20167473
- [Background] Tanaka JW, Sung A. The "Eye Avoidance" Hypothesis of Autism Face Processing. J Autism Dev Disord. 2016 May;46(5):1538-52. doi: 10.1007/s10803-013-1976-7. PMID 24150885
- [Background] Wieckowski AT, White SW. Attention Modification to Attenuate Facial Emotion Recognition Deficits in Children with Autism: A Pilot Study. J Autism Dev Disord. 2020 Jan;50(1):30-41. doi: 10.1007/s10803-019-04223-6. PMID 31520245
- [Background] Ramdoss S, Machalicek W, Rispoli M, Mulloy A, Lang R, O'Reilly M. Computer-based interventions to improve social and emotional skills in individuals with autism spectrum disorders: a systematic review. Dev Neurorehabil. 2012;15(2):119-35. doi: 10.3109/17518423.2011.651655. PMID 22494084
- [Background] Kouo JL, Egel AL. The Effectiveness of Interventions in Teaching Emotion Recognition to Children with Autism Spectrum Disorder. Rev J Autism Dev Disord. 2016 Sep;3(3):254-65.
- [Background] Silver M, Oakes P. Evaluation of a new computer intervention to teach people with autism or Asperger syndrome to recognize and predict emotions in others. Autism. 2001 Sep;5(3):299-316. doi: 10.1177/1362361301005003007. PMID 11708589
- [Background] Zoerner D, Schutze J, Kirst S, Dziobek I, Lucke U. Zirkus Empathico: Mobile Training of Socio-Emotional Competences for Children with Autism. In: 2016 IEEE 16th International Conference on Advanced Learning Technologies (ICALT) [Internet]. Austin, TX, USA: IEEE; 2016 [cited 2021 Feb 10]. p. 448-52. Available from: http://ieeexplore.ieee.org/document/7757020/
- [Background] Hunnikin LM, van Goozen SHM. How can we use knowledge about the neurobiology of emotion recognition in practice? Journal of Criminal Justice. 2019 Nov;65:101537.
- [Background] Cooper S, Hobson CW, van Goozen SH. Facial emotion recognition in children with externalising behaviours: A systematic review. Clin Child Psychol Psychiatry. 2020 Oct;25(4):1068-1085. doi: 10.1177/1359104520945390. Epub 2020 Jul 25. PMID 32713184
- [Background] Wells AE, Hunnikin LM, Ash DP, van Goozen SHM. Improving emotion recognition is associated with subsequent mental health and well-being in children with severe behavioural problems. Eur Child Adolesc Psychiatry. 2021 Nov;30(11):1769-1777. doi: 10.1007/s00787-020-01652-y. Epub 2020 Sep 30. PMID 32997168
- [Background] Dadds MR, Cauchi AJ, Wimalaweera S, Hawes DJ, Brennan J. Outcomes, moderators, and mediators of empathic-emotion recognition training for complex conduct problems in childhood. Psychiatry Res. 2012 Oct 30;199(3):201-7. doi: 10.1016/j.psychres.2012.04.033. Epub 2012 Jun 15. PMID 22703720
- [Background] Hubble K, Bowen KL, Moore SC, van Goozen SH. Improving Negative Emotion Recognition in Young Offenders Reduces Subsequent Crime. PLoS One. 2015 Jun 29;10(6):e0132035. doi: 10.1371/journal.pone.0132035. eCollection 2015. PMID 26121148
- [Background] Moebert, T. & Lucke, U., (2019). E.V.A. - Emotionen Verstehen und Ausdrücken. In: Pinkwart, N. & Konert, J. (Hrsg.), DELFI 2019. Bonn: Gesellschaft für Informatik e.V.. (S. 289-290). DOI: 10.18420/delfi2019_324
- [Background] Schlegel K, Grandjean D, Scherer KR. Introducing the Geneva emotion recognition test: an example of Rasch-based test development. Psychol Assess. 2014 Jun;26(2):666-72. doi: 10.1037/a0035246. Epub 2013 Dec 2. PMID 24295238